CLINICAL TRIAL: NCT03066622
Title: Oral Rapidly Dissolving Olanzapine for Acute Primary Headache in the Emergency Department Setting: A Feasibility Trial
Brief Title: Olanzapine for Acute Headaches
Acronym: Olanzapine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-420
Record Dates: First submitted 2016-12-06; First posted 2017-02-28 (Actual); Results first posted 2019-08-20 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2018-06

CONDITIONS: Headache
MeSH Terms: conditions — Headache | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, convenience sample, feasibility trial to test for non-inferiority of oral rapidly dissolving olanzapine versus current emergency department standard of care in providing symptomatic relief to patients presenting with primary headache.
Masking Description: Open label, not blinded, randomized 2-arm trial
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (Active Comparator): IV Morphine or any medication per attending decision
  Interventions: Drug: Standard of Care as per attending physician
- Olanzapine (Experimental): oral rapidly dissolving olanzapine (Zydis) 5 mg for analgesia in acute primary headaches.
  Interventions: Drug: 5mg rapidly dissolving olanzapine

INTERVENTIONS:
Drug: Standard of Care as per attending physician — Patients are randomized to standard of care medication (as determined by attending physician)
  Other Names: standard of care
  Arms: Standard of Care
Drug: 5mg rapidly dissolving olanzapine — 5mg rapidly dissolving olanzapine
  Other Names: Zydis
  Arms: Olanzapine

SUMMARY:
This trial is a prospective, randomized, feasibility trial with the primary aim of comparing how well oral rapidly dissolving olanzapine controls primary headache pain when compared to the current treatment strategies used in emergency departments which often require intravenous or intramuscular medications.

DETAILED DESCRIPTION:
Primary Question:

Does oral rapidly dissolving olanzapine provide efficacious analgesia in patients with acute headache of non-organic origin (primary headache) who come to the ED for abortive therapy when compared to current standard of care?

Secondary Aim:

Additionally, the study will aim to see if oral rapidly dissolving olanzapine decreases 1) duration of ED length of stay and 2) need for IV access when compared to the current standard of care.

This is a prospective, randomized, convenience sample, feasibility trial to test for non-inferiority of oral rapidly dissolving olanzapine versus current emergency department standard of care in providing symptomatic relief to patients presenting with primary headache.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient between 18-65 years of age presenting to the emergency department with acute primary headache
2. Patient approved for inclusion by primary attending physician in the emergency department

Exclusion Criteria:

1. Age < 18 or > 65
2. Pregnancy
3. Known allergy to olanzapine
4. Known QT prolongation or underlying condition that places patient at risk for QT prolongation
5. Inability to give written consent (intoxication, altered mental status)
6. Headache of organic origin (trauma, infection, previous recent head or neck surgery)
7. Patient already prescribed daily olanzapine on an outpatient basis
8. Patient has been administered olanzapine within the past 24 hours
9. Language barrier

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2018-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Hernandez, MD, Principal Investigator — HealthPartners Institute
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Standard of Care medication for treatment of headache as per attending physician: Patients are randomized to standard of care medication (as determined by attending physician)
Period: Overall Study
Arm/Group | Standard of Care | Olanzapine
Started | 61 | 61
Completed | 35 | 35
Not Completed | 26 | 26
Not completed — Lost to Follow-up | 24 | 25
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: The baseline population included is 119 as 5 subjects withdrew after providing informed consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Olanzapine | Total
Number analyzed (Participants) | 60 | 59 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (11.2) | 34.2 (10.5) | 34.2 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 42 | 89
  Male | 13 | 17 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 57 | 53 | 110
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 22 | 49
  White | 29 | 28 | 57
  More than one race | 2 | 6 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 60 | 59 | 119

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Scores Based on Patient Questionnaire
Description: Change in patient reported pain score from baseline using the Numeric Pain Rating Scale (PNRS) Minimum score = 0 Maximum score = 10 Lower score indicates lower pain level, with zero indicating no pain and 10 indicating the worst pain imaginable.
Time Frame: baseline, 30, 60, and 90 minutes post drug administration
Population: Not all participants were assessed at each time point due to some being discharged from the Emergency Department prior to study data collection time points.
Measure: Mean (Standard Deviation); unit: units on a scale of 1-10
Arm/Group | Standard of Care | Olanzapine
Number analyzed (Participants) | 58 | 56
units on a scale of 1-10
  Pain at 30 minutes | -2.95 (2.5) | -1.79 (1.83)
  Pain at 60 minutes: number analyzed (Participants) | 53 | 49
  Pain at 60 minutes | -4.49 (2.95) | -2.65 (2.36)
  Pain at 90 minutes: number analyzed (Participants) | 34 | 40
  Pain at 90 minutes | -4.68 (2.64) | -3.88 (2.79)

2. Secondary Outcome: Comparison of Duration of ED Length of Stay
Description: The total time the patient spent in the ED after initially being seen by the physician
Time Frame: Length of Emergency Department stay (Time Frame: up to 12 hours)
Population: Data was only available for 60 subjects in the standard of care arm and 58 subjects in the olanzapine arm.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Standard of Care | Olanzapine
Number analyzed (Participants) | 60 | 58
Minutes | 179.57 (83.67) | 180.28 (78.60)

3. Secondary Outcome: Number of Participants That Receive Peripheral Intravenous Catheterization
Description: Determining if patients randomized to rapidly dissolving Olanzapine eventually require IV access, defined as A successful cannulation (blood return or ability to infuse intravenous fluid without infiltration) on initial percutaneous needle puncture
Time Frame: Length of Emergency Department stay (Time Frame: up to 12 hours)
Population: Subjects consenting to participate in the study through time of ED discharge with complete data.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Olanzapine
Number analyzed (Participants) | 60 | 58
Participants | 55 | 28

ADVERSE EVENTS:
Time Frame: Adverse event data were collected until completion of the 48 hour follow-up phone call (24-72 hours following enrollment).
Arm/Group | Standard of Care | Olanzapine
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/59
Other Adverse Events (participants affected / at risk) | 12/60 | 11/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=60) | Olanzapine (N=59)
Dizziness, lightheadedness (General disorders) | 4 (4) | 2 (2)
Drowsiness (General disorders) | 2 (2) | 6 (6)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Burning sensation at IV site (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ringing in ears (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Jittery feeling (General disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT03066622/Prot_SAP_000.pdf